CLINICAL TRIAL: NCT04946552
Title: Sympathetic Activation in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000030749; 1R56DK129344-01 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-07-01 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Healthy
MeSH Terms: conditions — Obesity | interventions — Positron-Emission Tomography; Glucose Tolerance Test; Body Composition; Tomography, X-Ray Computed; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with normal BMI (Active Comparator): (BMI 18-25 kg/m2)
  Interventions: Diagnostic Test: PET Scan; Dietary Supplement: Mixed Meal Test; Diagnostic Test: Muscle sympathetic nerve activity (MSNA); Diagnostic Test: Oral Glucose Tolerance Test; Other: Body Composition, Percent Body Fat & Percent Body Water (Tanita scale); Diagnostic Test: CT Scan; Other: Body Composition, Percent Body Fat & Percent Body Water (DXA Scan)
- Individuals with obesity (Active Comparator): (BMI 30-40 kg/m2)
  Interventions: Diagnostic Test: PET Scan; Dietary Supplement: Mixed Meal Test; Diagnostic Test: Muscle sympathetic nerve activity (MSNA); Diagnostic Test: Oral Glucose Tolerance Test; Other: Body Composition, Percent Body Fat & Percent Body Water (Tanita scale); Diagnostic Test: CT Scan; Other: Body Composition, Percent Body Fat & Percent Body Water (DXA Scan)

INTERVENTIONS:
Diagnostic Test: PET Scan — Participants will come to the PET Center to undergo the whole body [11C]MRB PET scan. An intravenous bolus dose of MRB (~20mCi) will be injected by an infusion pump. PET data will be acquired dynamically for 120 min using the Siemens mCT-X whole-body PET/CT scanner using continuous bed motion to image multiple PET bed acquisitions from the top of the head to the lower abdominal region.
Dietary Supplement: Mixed Meal Test — High Carbohydrate Mixed Meal Test (MMT): participants will be studied after a 10-hour overnight fast. A nurse will insert an intravenous (IV) catheter and subjects will ingest a liquid meal (65% carbohydrate, 20% fat, and 15% protein, corresponding to 40% of daily energy expenditure, in ~16 ounces) to be prepared by the Hospital Research Unit Metabolic Kitchen. Blood samples will be collected at -10, 0, 15, 30, 60, 90, and 120 min) for measurement of glucose, insulin and C-peptide concentrations. Plasma samples will be drawn at baseline and throughout the MMT for measurement of additional hormones (such as thyroid hormones, and catecholamines) and free fatty acids (FFA) levels.
Diagnostic Test: Muscle sympathetic nerve activity (MSNA) — Recording of multiunit postganglionic muscle sympathetic nerve activity (MSNA) will be made from the common peroneal nerve as it winds around the fibular head with the subject in the supine position with the subject's thigh comfortably supported. This procedure requires to first trace the course of the nerve using small electrical stimuli applied to the surface of the skin over the nerve or use of ultrasound to visually assist.
Diagnostic Test: Oral Glucose Tolerance Test — Following a 10-hour overnight fast, a nurse will insert an intravenous (IV) catheter. Subsequently, subjects will ingest 7.5 oz of Glucola, which contains 75 g of dextrose in orange flavored water. Blood samples will be taken at -15, 0, 10, 20, 30, 60, 90 and 120 minutes (after glucola ingestion) for the measurement of plasma glucose, insulin, and C-peptide concentrations, and calculation of measurements of insulin sensitivity index (Matsuda Index). Approximately 40 mL of blood will be drawn at this visit.
Other: Body Composition, Percent Body Fat & Percent Body Water (Tanita scale) — will be assessed using bioelectrical impedance analysis Tanita® scale; which is a special multi frequency segmental body composition analyzer that delivers a very mild electrical current that allows measurement of fat mass, percent body fat, fat free mass, total body water, and percent body water. This test will be performed at screening visit.
Diagnostic Test: CT Scan — A CT scan will be performed for attenuation correction and to help delineate the BAT and other regions of interest (ROIs). Images will be reconstructed with an ordered subset expectation maximization algorithm using point spread function correction and time-of-flight information. To delineate fat (WAT, BAT) and skeletal muscle regions of interests (ROIs), CT images are first resliced to match the resolution and location of PET images. As performed in previous studies 2, a supraclavicular ROI is first manually drawn on the CT images. Within that area, the fat ROI is segmented using the CT images and an intensity window from -200 to -50 HU. Subsequently the fat ROI is segmented into WAT and BAT ROIs by using the 11C-MRB PET images: Standardized Uptake Value (SUV) ≥ 1.25 for BAT, SUV < 1.25 for WAT.
Other: Body Composition, Percent Body Fat & Percent Body Water (DXA Scan) — For better accuracy, measurement of percent fat and percent body water will be obtained with whole body Dual X-Ray Absorptiometry (DXA) scan (Hologic®) on screening-OGTT visit. The scanner arm will move over the participant's body from feet to head. The machine uses a small amount of radiation (one tenth of the amount of radiation from a chest x-ray) to measure body fat, muscle and bone density.

SUMMARY:
The primary objective of this study is to determine whether sympathetic nervous system (SNS) activity in white adipose tissue (WAT) and brown adipose tissue (BAT), skeletal muscle and brain is altered in individuals with obesity in comparison to individuals with normal weight. Simultaneous multi-organ SNS activation will be obtained with a radiotracer for norepinephrine transporter (NET) for whole-body Positron Emission Tomography (PET) imaging and microneurography (peroneal muscle SNS activity).

The secondary objectives of this study are: 1) to evaluate whether gender differences affect peripheral SNS in healthy normal weight and obese men and women in adipose tissue (WAT and BAT) and muscle (resting/fasting); 2) To investigate the relationship between peripheral and central SNS activity in obesity, by correlating SNS activity in peripheral tissues (WAT, BAT, and muscle) and brain; and 3) To investigate NET CNS and peripheral SNS activity before and after a high carbohydrate mixed meal in lean and obese men and women.

ELIGIBILITY:
Inclusion Criteria:In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age 18-45 years
4. In good general health as evidenced by medical history and lean (BMI 18.5-24.9 kg/m2) or non-diabetic obese (BMI 30-50 kg/m2) with a fasting plasma glucose (FPG) <100 mg/dL and a hemoglobin A1c <5.7%.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Hypertension
2. Cardiac or pulmonary disease,
3. Known history of Type 1 or Type 2 diabetes
4. Hepatic disease, swallowing and gastrointestinal disorders
5. Current use of anti-obesity medications, supplements and/or anti-hyperglycemic medications
6. Neurological injury or illness, and psychiatric medications
7. Women who are pregnant or lactating
8. Subjects who suffer from claustrophobia
9. Subjects who have received a diagnostic or therapeutic radiopharmaceutical within 7 days prior to participation in this study
10. Radiation works or participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the subject to exceed the yearly dose limits.
11. Subjects with history of IV drug use which would prevent venous access for PET tracer injection
12. Severe motor problems that prevent the subject from lying still for PET and MR imaging
13. Subjects who complain of chronic pain
14. Blood donation within 8 weeks of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Church Street Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Individuals With Normal BMI: BMI 18-25 kg/m2 PET Scan, Mixed Meal Test, Muscle sympathetic nerve activity (MSNA), Oral Glucose Tolerance Test, Body Composition, Percent Body Fat & Percent Body Water, CT Scan
- Individuals With Obesity: BMI 30-40 kg/m2 PET Scan, Mixed Meal Test, Muscle sympathetic nerve activity (MSNA), Oral Glucose Tolerance Test, Body Composition, Percent Body Fat & Percent Body Water, CT Scan
Period: Overall Study
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Presented are baseline characteristics across both arms to preserve anonymity.
Groups:
- Overall: Presented are baseline characteristics overall as there were only 2 people in a single treatment arm and therefore identifying information could be obtained.
Arm/Group | Overall
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 2
  White | 3
Region of Enrollment [Number; unit: participants]
  United States | 5
Weight [Mean (Standard Deviation); unit: kilograms] | 68.45 (4.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.65 (2.5)
Systolic Blood Pressure (BP) [Mean (Standard Deviation); unit: mmHg] | 108.85 (8.55)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 67.85 (6.6)
Insulin Sensitivity Index (ISI) Score using the Matsuda Index [Mean (Standard Deviation); unit: score on a scale] — An assessment of insulin sensitivity that provides a reasonable approximation of whole-body insulin sensitivity. Insulin sensitivity was calculated with Matsuda index: [10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT)]. Scores range from 0-12 with higher scores indicating better insulin sensitivity.
  score on a scale | 2.95 (0.65)
Study Group [Count of Participants; unit: Participants]
  Obese Group (BMI Greater than 25 kg/m2) | 2
  Lean Group (BMI 18-25 kg/m2) | 3

OUTCOME MEASURES:

1. Primary Outcome: Distribution Volume Ratio (DVR) of [11C]MRB PET Imaging of Peripheral Sympathetic Nervous System
Description: Lean individuals with a BMI of 18-25 and obese individuals with a BMI of 30-40 will undergo a PET/CT scan to determine group differences in sympathetic nervous system (SNS) activity in white adipose tissue (WAT), brown adipose tissue (BAT), and deltoid muscle. SNS activity will be determined by using [11C]MRB a radiotracer for PET imaging.
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: DVR
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
DVR
  Brain: Putamen | 0.13 (0.014) | -0.025 (0.120)
  Brain: Caudate | 0.095 (0.063) | -0.03 (0.028)
  Brain: Hypothalamus | -0.095 (0.691) | -0.195 (0.332)
  Brain: Locus Ceruleus | -1.47 (1.49) | -0.01 (0.283)
  Brain: Thalamus | 0.295 (0.205) | -0.115 (0.092)
  Brain: Raphe | -0.255 (0.049) | -0.455 (0.657)
  Brain: Paracentral Lobule | 0.045 (0.587) | -0.055 (0.191)
  Muscle: Deltoid | 0.525 (0.058) | 0.549 (0.107)

2. Primary Outcome: Microneurography (Muscle Sympathetic Nerve Activity (MSNA)) Measured by Burst Frequency
Description: Muscle sympathetic nerve activity will be quantified by identification and measurement of sympathetic bursts in the integrated neurogram and expressed as burst frequency (mean number of bursts per unit time) to determinate group differences in peroneal MSNA at baseline (fasting) and during MMT.
Time Frame: 30-60 minutes
Measure: Mean (Standard Deviation); unit: bursts per minute
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
bursts per minute
  Fasting | 11.18 (1.58) | 9.541 (0.245)
  MMT | 15.63 (4.8) | 11.60 (2.61)

3. Secondary Outcome: DVR of Norepinephrine Transporter (NET) in the Central Nervous System (CNS)
Description: Regional quantification of [11C]MRB uptake as distribution volume ratio (DVR ) will be used to measure NET in the CNS.
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: DVR
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
DVR | 0.549 (0.107) | 0.525 (0.058)

4. Secondary Outcome: DVR of [11C]MRB PET Imaging of Peripheral Sympathetic Nervous System After Mixed Meal Test
Description: Measurement of peripheral SNS Activity with [11C]MRC for PET/CT before (fasting) and after a high carbohydrate mixed meal in individuals with normal weight and obesity.
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: DVR
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
DVR
  Fasting | 0.577 (0.121) | 0.491 (0.041)
  MMT | 0.521 (0.128) | 0.559 (0.061)

5. Secondary Outcome: Plasma Glucose
Description: Measurement of plasma glucose levels will be obtained at fasting and during the Mixed Meal Test (MMT). The normal range for glucose levels is 70-100 mg/dL.
Time Frame: 2 hours
Population: Data for this outcome was not collected
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Insulin Levels
Description: Measurement of plasma insulin levels will be obtained at fasting and during the MMT. Insulin levels in the plasma are higher in individuals with obesity. The normal range for insulin is: < or = 19.6 mcg/dL
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
uU/mL
  Fasting | 7.07 (0.568) | 15.55 (0.327)
  MMT | 61.06 (54.3) | 78.37 (45.96)

7. Secondary Outcome: C-Peptide
Description: Plasma samples will be drawn at baseline and throughout the MMT for measurement of C-Peptide. The normal range for C-Peptide is 0.80 - 3.85 ng/mL
Time Frame: 2 hours
Population: Data for this outcome was not collected
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Plasma Catecholamines (Epinephrine and Norepinephrine)
Description: Measurement of epinephrine and norepinephrine levels in the plasma at fasting and during the MMT. The normal range for epinephrine is 0 to 140 pg/mL (764.3 pmol/L). The normal range for norepinephrine is 70 to 1700 pg/mL (413.8 to 10048.7 pmol/L).
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
mg/mL
  Epinephrine Fasting | 0.0487 (0.0167) | 0.0131 (0.0238)
  Epinephrine MMT | 0.0155 (0) | 0.0136 (0.0138)
  Norepinephrine Fasting | 0.146 (0.0376) | 0.135 (0.0572)
  Norepinephrine MMT | 0.278 (0.109) | 0.162 (0.0779)

9. Secondary Outcome: Plasma Free Fatty Acids (FFA)
Description: Percent of plasma free fatty acids levels will be obtained at fasting and during the Mixed Meal Test (MMT). FFA levels in the plasma are higher in individuals with obesity than individuals with normal weight.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percentage of FFA
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
percentage of FFA
  Fasting | 380 (42.91) | 412 (37.702)
  MMT | 419 (19.20) | 404 (35.40)

10. Secondary Outcome: Thyroid Function Tests
Description: Plasma samples will be drawn at baseline and throughout the mixed meal test (MMT) for measurement of Thyroid Stimulating Hormone (TSH), free T4 (FT4) and total T3 (TT3). The normal range for TSH is : 0.4-4.5 mlU/L, FT4: 0.8-1.8 ng/dL, TT3: 76 - 181 ng/dL.
Time Frame: 2 hours
Population: Data for this outcome was not collected
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Electrocardiogram (EKG)- Heart Rate
Description: EKG surface electrodes will be applied to the chest for measurement of heart rate and heart rate variability (QT Interval).
Time Frame: 30-60 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
beats per minute
  Fasting | 61.8 (6.47) | 74.2 (4.06)
  MMT | 65.6 (9.97) | 71.7 (5.32)

12. Secondary Outcome: Electrocardiogram (EKG) - RR Interval
Description: EKG surface electrodes will be applied to the chest for measurement of RR interval.
Time Frame: 30-60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
Number analyzed (Participants) | 3 | 2
seconds
  Fasting | 0.94 (0.16) | 1.01 (0.11)
  MMT | 0.91 (0.07) | 0.85 (0.16)

ADVERSE EVENTS:
Time Frame: Up to 120 minutes
Arm/Group | Individuals With Normal BMI | Individuals With Obesity
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04946552/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04946552/ICF_001.pdf